CLINICAL TRIAL: NCT05343819
Title: A Randomized, Single-center, Double-blind, Placebo Controlled Trial With Ascending Multiple Intravenous Doses to Determine Safety, Tolerability and Pharmacokinetics of AON-D21 in Healthy Male Subjects.
Brief Title: Ascending Multiple Intravenous Doses of AON-D21 in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptarion Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-D21-C200; 2021-006551-33 (EudraCT Number)
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Sequential: Two groups of participants will be assigned to receive AON-D21 or placebo in ascending dose order. Dose will be escalated based on safety and pharmacokinetic data.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: Participant, Investigator, Outcomes Assessor and Care provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AON-D21 (Experimental): Multiple ascending doses by iv infusion
  Interventions: Drug: AON-D21
- Placebo (Placebo Comparator): Placebo medication identical in appearance to active
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AON-D21 — AON-D21 is a PEGylated L-configured aptamer that binds and thereby neutralizes the complement component C5a from activating both C5a receptors.
  Arms: AON-D21
Drug: Placebo — Isotonic glucose solution identical in appearance to AON-D21.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamic parameters after multiple ascending intravenous doses of AON-D21 in healthy male subjects.

DETAILED DESCRIPTION:
This study will potentially include 2 two sequential cohorts with 8 healthy male subjects per cohort, then 16 enrolled subjects in total. Within each dose group 6 subjects will be randomized to receive AON-D21 and 2 subjects will be randomly assigned to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Body mass index (BMI) within the range 18 - 30 kg/m2 with a body weight between 50 kg and 120 kg.
* Male subjects
* Subject is healthy as determined by medical evaluation
* Subject provided written informed consent
* Subject is willing to comply with all requirements and restrictions according to the study protocol.

Exclusion Criteria:

* Any concomitant disease, condition, or treatment that could interfere with the conduct of the study.
* Any acquired or congenital immune deficiency.
* Acute infection (including viral infections) in the preceding 6 weeks (8 weeks for respiratory infections).
* Clinically relevant abnormality following the Investigator's review of the physical examination, vital signs, ECG and clinical study protocol-defined clinical laboratory tests that, in the opinion of the Investigator, would preclude inclusion in the trial at screening and admission.
* Evidence of COVID-19 signs or symptoms, exposure to infected person or confirmed COVID-19 infection within the last 2 weeks.
* Use of any concomitant medication or prescribed or non-prescribed drugs within 2 weeks or 5 times the half-life, whichever is longer, prior to the first study treatment administration.
* Administration of vaccine(s) within 2 weeks prior to screening or plans to receive such vaccines during the study.
* Use of any investigational drug or participation in any clinical study within 30 days or 5 half-life times, whichever is longer, prior to dosing.
* Positive drug or alcohol screen at screening and admission.
* Any significant blood loss, donated one unit (450 mL) of blood or more, or donated plasma, or received a transfusion of any blood or blood products within 30 days prior to dosing.
* Subjects who are unable to refrain from the consumption of Seville oranges, grapefruit or grapefruit juice and /or pomelos, exotic citrus fruits, grapefruit hybrids, starfruit or fruit juices from 72 hours prior to dosing on Day 1, until completion of the last PK blood sample time point.
* Legal incapacity or limited legal capacity, or incarceration.
* Inability to understand or communicate reliably with the Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 27 days
  Nature, occurrence, and severity of treatment-emergent adverse events.
Per dosing cohort number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0. | 27 days
  Overall number of participants with treatment related treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0 per dosing cohort.

SECONDARY OUTCOMES:
Pharmacokinetics assessment | 27 days
  Area under the concentration-time curve (AUC) over the dosing interval at steady state (AUC0-tau) of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Maximum concentration at steady state (Cmax) of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Average drug concentration at steady state (Cav) of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Trough concentrations (Ctrough) of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Time of maximum concentration at steady state (Tmax) of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Terminal half-life at steady state (t1/2) of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Accumulation ratios for Cmax and AUC of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Clearance (CL) of AON-D21 in plasma at steady state.
Pharmacokinetics assessment | 27 days
  Volume of distribution (Vz) of AON-D21 in plasma at steady state.
Pharmacokinetics assessment | 27 days
  AUC from 0 to 48 hours (AUC0-48) after the first dose of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  AUC from 0 extrapolated to infinity (AUC0-inf) after the first dose of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Maximum concentration (Cmax) after the first dose of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Time to maximum concentration (Tmax) after the first dose of AON-D21 in plasma.
Pharmacokinetics assessment | 27 days
  Terminal half life (t1/2) after the first dose of AON-D21 in plasma.
Pharmacodynamics assessment | 27 days
  Measurement of concentration of C5 in plasma.
Pharmacodynamics assessment | 27 days
  Measurement of concentration of C5a in plasma.
Pharmacodynamics assessment | 27 days
  Measurement of concentration of C5b-9 in plasma.
Pharmacodynamics assessment | 27 days
  Qualitative assessment of terminal complement complex (TCC) formation in plasma.
To assess potential for immunogenicity | 27 days
  Measurement of anti-drug antibodies (ADA) in plasma.
To assess potential for immunogenicity | 27 days
  Measurement of anti-polyethylene glycol (PEG) antibodies in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Koch, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No